CLINICAL TRIAL: NCT04452214
Title: An Open-label, Safety and Tolerability Phase 1b Trial of CAN04, a Fully Humanized Anti-IL1RAP Monoclonal Antibody, and Pembrolizumab in Combination With and Without Carboplatin and Pemetrexed in Subjects With Solid Tumors
Brief Title: A Study of the Safety and Tolerance of CAN04 and Pembrolizumab in Combination With and Without Carboplatin and Pemetrexed in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cantargia AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN04CLIN002
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Urothelial Carcinoma; Malignant Melanoma; Head and Neck Squamous Cell Carcinoma
Keywords: NSCLC; Adenocarcinoma of lung; Lung cancer; Squamous cell lung cancer; Malignant melanoma; Urothelial cancer; Non-small-cell lung cancer; Non small cell lung cancer; Non-small-cell lung carcinoma; Non small cell lung carcinoma; HNSCC; Head and neck squamous cell carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Melanoma; Squamous Cell Carcinoma of Head and Neck; Adenocarcinoma of Lung; Lung Neoplasms | interventions — pembrolizumab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAN04 and pembrolizumab (Part 1) (Experimental): Subjects will receive weekly doses of CAN04 in combination with pembrolizumab given as standard regimen
  Interventions: Drug: CAN04; Drug: Pembrolizumab
- CAN04 + pembrolizumab + carboplatin + pemetrexed (Part 2) (Experimental): Subjects will receive doses of CAN04 on Days 1 and 8 (Cycles 1 thru 4), and on Day 1 (Cycle 5 onwards) in combination with pembrolizumab given as standard regimen and carboplatin and pemetrexed standard of care
  Interventions: Drug: CAN04; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: CAN04 — Administered intravenously
Drug: Pembrolizumab — Administered intravenously
Drug: Carboplatin — Administered intravenously
  Arms: CAN04 + pembrolizumab + carboplatin + pemetrexed (Part 2)
Drug: Pemetrexed — Administered intravenously
  Arms: CAN04 + pembrolizumab + carboplatin + pemetrexed (Part 2)

SUMMARY:
This study will consider the safety and effectiveness of a study drug, CAN04, in combination with pembrolizumab, in the treatment of incurable or metastatic non-small-cell lung cancer (NSCLC), head and neck squamous cell carcinoma, urothelial cancer, or malignant melanoma. The study aims to establish a recommended dose of CAN04 in combination with the standard dose of pembrolizumab (Part 1), and in combination with pembrolizumab standard dose, and Standard of Care carboplatin and pemetrexed (Part 2 - subjects with stage IV, non-squamous metastatic NSCLC). CAN04, pembrolizumab. carboplatin and pemetrexed will be administered intravenously.

ELIGIBILITY:
Inclusion Criteria (Part 1):

* Subjects with metastatic or locally advanced, incurable non-small-cell lung cancer (NSCLC [adenocarcinoma, adenosquamous, or squamous]), head and neck squamous cell carcinoma (HNSCC), urothelial cancer, or malignant melanoma who have exhausted or declined available standard therapy.
* Subjects progressing on previous treatment with a checkpoint inhibitor targeting thePD-1/PD-L1 pathway, alone or in combination with chemotherapy after previously having achieved stable disease or better and stayed on such therapy for ≥12 weeks.
* Primary or metastatic lesion suitable for biopsy and willingness to undergo repeat biopsies as appropriate.
* Willing and able to provide intravenous access for the administration of the study drug and for blood sampling/testing.

Inclusion Criteria (Part 2):

* Subjects with histologically confirmed non-squamous metastatic (stage IV) NSCLC, without option for locoregional treatment with curative intent.
* Subjects who have not received prior systemic anti-cancer therapy for the locally advanced or metastatic NSCLC. Subjects who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of metastatic disease.
* Ability to safety undergo pre-treatment (if no archival biopsy is available) and on-treatment tumor biopsies.
* Subject consents to retrieval of archival tumor tissue for screening in case no fresh biopsy is performed during screening.
* Willing and able to provide intravenous access for the administration of the study drug and for blood sampling/testing.

Exclusion Criteria (Parts 1 and 2):

* Subjects with NSCLC tumors with genetic alteration or mutation, for which FDA-approved targeted therapy is available.
* Treatment with systemic anticancer treatments, investigational products, or major surgery within 4 weeks before first dose of study drug or 5 half-lives, whichever is shorter. Subjects should have recovered from previous treatment toxicity (except hair loss and peripheral neuropathy).
* History of uncontrolled brain metastasis.
* Subject has received extended field radiotherapy ≤4 weeks before the start of treatment (≤2 weeks for limited field radiation to alleviate symptoms), and who has not recovered from related side effects of such therapy (except for hair loss).
* Subjects who have previously experienced an immune-related adverse event (irAE) to pembrolizumab, for which permanent discontinuation is required. Subjects without a formal contraindication due to previous irAE are not eligible if the AE has not resolved or requires steroids (>10 mg prednisone-equivalent per day) for ongoing management.
* Subjects with active severe infection requiring oral antibiotics.
* Clinical evidence of an active second invasive malignancy with the exception of stable prostate cancer on watchful waiting.
* Uncontrolled or significant cardiovascular disease.
* History of autoimmune disease requiring systemic immunosuppressive therapy (daily prednisone equivalent doses >10 mg/day).
* HIV patients can be enrolled if the infection is adequately controlled.
* Known bleeding disorder or coagulopathy. Subjects on stable anticoagulant therapy are allowed.
* Known or suspected allergy to study treatment or related products.
* Women who are pregnant or breastfeeding, or trying to become pregnant.
* Patients with chronic viral hepatitis.

Exclusion criteria (Part 2):

* Previous therapy with immunotherapy (anti-PD-1, anti-PD-L1, and anti-PD-L2, anti-CTLA-4, or other approved or investigational checkpoint-inhibitors).
* Subject is unable or unwilling to take folic acid or vitamin B12 supplementation.
* Subject is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDS), other than an aspirin dose ≤ 1.3 g per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Frequency of TEAEs (treatment-emergent adverse events) (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Frequency of TEAEs (treatment-emergent adverse events) (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Number of participants with DLTs (dose-limiting toxicities) (Part 1) | Up to day 28
Number of participants with DLTs (dose-limiting toxicities) (Part 2) | Up to day 28
Number of subjects with grade ≥3 TEAEs (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Number of subjects with grade ≥3 TEAEs (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Percentage of subjects with grade ≥3 TEAEs (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Percentage of subjects with grade ≥3 TEAEs (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Number of subjects with 1 or more SAEs (serious adverse events) (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Number of subjects with 1 or more SAEs (serious adverse events) (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Percentage of subjects with 1 or more SAEs (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Percentage of subjects with 1 or more SAEs (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Number of subjects with 1 or more TEAEs leading to dose modifications (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Number of subjects with 1 or more TEAEs leading to dose modifications (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Number of subjects with 1 or more TEAEs leading to treatment discontinuation (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Number of subjects with 1 or more TEAEs leading to treatment discontinuation (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Percentage of subjects with 1 or more TEAEs leading to dose modifications (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Percentage of subjects with 1 or more TEAEs leading to dose modifications (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Percentage of subjects with 1 or more TEAEs leading to treatment discontinuation (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Percentage of subjects with 1 or more TEAEs leading to treatment discontinuation (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first

SECONDARY OUTCOMES:
Serum concentrations of CAN04 and pembrolizumab (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Serum concentrations of CAN04 and pembrolizumab (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Antidrug antibodies (ADAs) against CAN04 | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Change in serum IL-6 (interleukin-6) concentration (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Change in serum IL-6 (interleukin-6) concentration (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Change in serum CRP (C-reactive protein) concentration (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Change in serum CRP (C-reactive protein) concentration (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Overall response rate (ORR) (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
  Proportion of subjects with partial response (PR) or complete response (CR) to study treatment as defined by iRECIST (immune-related response evaluation criteria in solid tumors) and measured by radiological assessment (CT/MRI scan)
Overall response rate (ORR) (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
  Proportion of subjects with partial response (PR) or complete response (CR) to study treatment as defined by iRECIST (immune-related response evaluation criteria in solid tumors) and measured by radiological assessment (CT/MRI scan)
Progression free survival (Part 1) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Progression free survival (Part 2) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first
Overall survival (Part 1) | Up to 36 months after 1st dose of last subject (or death)
Overall survival (Part 2) | Up to 36 months after 1st dose of last subject (or death)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Garcia-Ribas, MD, PhD, Study Director — Cantargia AB
Locations (3):
- United States (3):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Florida Cancer Specialists & Research Institute, Lake Mary, Florida
  - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: FDA Recalls, Market Withdrawals, and Safety Alerts — http://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts